CLINICAL TRIAL: NCT01686087
Title: Attaining and Maintaining Wellness in OCD
Brief Title: Attaining and Maintaining Wellness in Obsessive-compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Helen Blair Simpson, Professor of Clinical Psychiatry, College of Physicians and Surgeons, Columbia University Director of the Anxiety Disorders Clinic and OCD Research Program, New York State Psychiatric Institute, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6628; 2R01MH045436-18 (NIH)
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuation of SRI (Active Comparator): Patients who achieve minimal to mild OCD symptoms and are not currently depressed at end of preparatory phase will be randomized to stay on SRI. They will receive 45 minute EX/RP booster sessions once per month.
  Interventions: Behavioral: Monthly Booster Sessions of EX/RP; Procedure: Visits with MD and independent evaluators
- Replace SRI w/placebo (Placebo Comparator): Patients who achieve minimal to mild OCD symptoms and are not currently depressed at end of preparatory phase will be randomized to gradual replacement with pill placebo. They will receive 45 minute EX/RP booster sessions once per month.
  Interventions: Behavioral: Monthly Booster Sessions of EX/RP; Procedure: Visits with MD and independent evaluators

INTERVENTIONS:
Behavioral: Monthly Booster Sessions of EX/RP — 45 minute EXRP booster sessions each month
Procedure: Visits with MD and independent evaluators — All patients will be followed carefully and evaluated by their study doctor and an independent evaluator to assess their symptoms.

SUMMARY:
The goal of this study is to understand whether patients with obsessive-compulsive disorder (OCD) on serotonin reuptake inhibitors (SRIs) who receive a type of Cognitive-behavioral therapy called Exposure and Ritual Prevention (EX/RP) can discontinue their medication if they first do well with EX/RP.

DETAILED DESCRIPTION:
This study begins with a Preparatory Phase, wherein all eligible participants receive up to 25 sessions of Exposure and Ritual Prevention (EX/RP) therapy. At the end of the Preparatory Phase, those who have achieved wellness (mild to minimal symptoms) enter the Study Phase. Those who do not achieve wellness will not continue in the study and are referred for treatment elsewhere. Those who enter the Study Phase are then assigned by chance to one of two groups. One group will continue on the SRI medication and the other group will discontinue the SRI gradually over 4-6 weeks as it is replaced with a placebo (sugar pill). Neither patients nor study staff will know which group a participant is in. Both groups will continue to receive monthly sessions of EX/RP. The study will examine who has the best response to treatment in this study, including taking blood samples for genetic testing to see whether there are genes that can predict who will or will not benefit from EX/RP.

ELIGIBILITY:
Preparatory Phase

Inclusion Criteria:

* Primary diagnosis of OCD
* Currently on a stable and adequate dose of a serotonin reuptake inhibitor (i.e., clomipramine, fluoxetine, fluvoxamine, sertraline, paroxetine, citalopram, escitalopram) but still have clinically significant OCD symptoms

Exclusion Criteria:

* Comorbid Psychiatric conditions that significantly elevate the risks of study participation (e.g. psychotic disorders, bipolar disorder, evidence of dementia or other cognitive disorder, suicidality)
* Unstable medical conditions that need attention and would make participation in the study unsafe (e.g., very high blood pressure)
* Patients who have already had prior adjunctive EX/RP (more than 8 sessions within 2 months) while receiving an adequate SRI trial
* Patients taking other medications besides an SRI (e.g. antipsychotics, mood stabilizers, other antidepressants besides SRIs)
* Patients who are pregnant, sexually active and not using contraception, or nursing

Study Phase

Inclusion Criteria:

* Those who achieve mild to minimum OCD symptoms from Preparatory Phase will enter the Study Phase

Exclusion Criteria:

* All exclusions listed above for Preparatory Phase are exclusions for Study Phase as well
* Patients who are depressed at the end of the Preparatory phase are excluded from Study Phase

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Obsessive Compulsive Symptom Severity (Y-BOCS) | 6 months
  In study phase, to determine whether those who have achieved wellness with Cognitive Behavioral Therapy who are on medication can maintain wellness when medication is stopped

SECONDARY OUTCOMES:
Depressive severity (HAMD17) | 6 months
  Hamilton Depression Scale (HAMD, 17 item)
Quality of Life (QLESQ-S) | 6 months
  Quality of Life Satisfaction Questionnaire (QLESQ, short form)

CONTACTS AND LOCATIONS:
Overall Officials: Helen B Simpson, MD PhD, Principal Investigator — NY State Psychiatric Institute at Columbia University; Edna Foa, PhD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - New York State Psychiatric Institute, New York, New York
  - University of Pennsylvania Center for the Treatment and Study of Anxiety, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Wheaton MG, Kalanthroff E, Mandel M, Marsh R, Simpson HB. Neurocognitive performance in obsessive-compulsive disorder before and after treatment with cognitive behavioral therapy. J Behav Ther Exp Psychiatry. 2025 Jun;87:102019. doi: 10.1016/j.jbtep.2025.102019. Epub 2025 Jan 20. PMID 39879875
- [Derived] Foa EB, Simpson HB, Gallagher T, Wheaton MG, Gershkovich M, Schmidt AB, Huppert JD, Imms P, Campeas RB, Cahill S, DiChiara C, Tsao SD, Puliafico A, Chazin D, Asnaani A, Moore K, Tyler J, Steinman SA, Sanches-LaCay A, Capaldi S, Snorrason I, Turk-Karan E, Vermes D, Kalanthroff E, Pinto A, Hamlett GE, Middleton R, Hahn CG, Xu B, Van Meter PE, Katechis M, Rosenfield D. Maintenance of Wellness in Patients With Obsessive-Compulsive Disorder Who Discontinue Medication After Exposure/Response Prevention Augmentation: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Mar 1;79(3):193-200. doi: 10.1001/jamapsychiatry.2021.3997. PMID 35080598